CLINICAL TRIAL: NCT02206763
Title: A Phase 1b Study of Erlotinib and Momelotinib for the Treatment of Epidermal Growth Factor Receptor (EGFR) Mutated EGFR Tyrosine Kinase Inhibitor (TKI) Naïve Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Erlotinib and Momelotinib for the Treatment of Epidermal Growth Factor Receptor (EGFR) Mutated EGFR Tyrosine Kinase Inhibitor (TKI) Naive Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-370-1298
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: EGFR Mutated EGFR TKI Naive Metastatic NSCLC
MeSH Terms: interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Momelotinib (MMB)+erlotinib (Experimental): Participants will receive momelotinib (MMB) plus erlotinib.
  Interventions: Drug: Momelotinib (MMB); Drug: Erlotinib

INTERVENTIONS:
Drug: Momelotinib (MMB) — Tablet(s) administered orally once or twice daily
  Other Names: GS-0387; CYT387
Drug: Erlotinib — Tablet(s) administered orally once daily.
  Other Names: Tarceva®

SUMMARY:
This study will evaluate the safety, preliminary efficacy, and pharmacokinetics (PK) of momelotinib (MMB) and erlotinib, as well as define the maximum tolerated dose (MTD) of momelotinib (MMB) combined with erlotinib in adults with epidermal growth factor receptor (EGFR)-mutated, EGFR tyrosine kinase inhibitor (TKI) naive metastatic non-small cell lung cancer (NSCLC). Participants will be sequentially enrolled to receive progressively increasing doses of momelotinib (MMB) in combination with erlotinib. Escalation of momelotinib (MMB) doses will proceed to the MTD, defined as the highest tested dose associated with dose-limiting toxicities (DLT) during the first 28 days of combined erlotinib and momelotinib (MMB) treatment. There will be four dose levels and each treatment cycle will consist of 28 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Metastatic NSCLC with documented EGFR exon 19 deletion or exon 21 (L858R) substitution mutation
* Treatment naive OR one prior standard chemotherapy that is platinum-based
* Adequate organ function defined as follows:

  * Hepatic: Total bilirubin < upper limit of the normal range (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
  * Hematological: absolute neutrophil count (ANC) ≥1500 cells/mm^3, platelet ≥ 100,000 cells/mm^3, hemoglobin ≥ 9.0 g/dL
  * Renal: Serum creatinine < ULN OR calculated creatinine clearance (CLcr) of ≥ 60 ml/min
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2

Key Exclusion Criteria:

* Known positive status for human immunodeficiency virus (HIV)
* Chronic active or acute viral hepatitis A, B, or C infection (testing required for hepatitis B and C)
* Presence of > Grade 1 peripheral neuropathy
* Symptomatic leptomeningeal, brain metastases, or spinal cord compression.
* History of interstitial pneumonitis

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose limiting toxicities refer to toxicities experienced during the first 28 days of combined erlotinib and momelotinib (MMB) treatment that have been judged to be clinically significant and related to study treatment.
Safety as Assessed by the Incidence of Adverse Events (AEs) | Up to 2 years plus 30 days
Safety as Assessed by the Percentage of Participants Experiencing Treatment-Emergent Graded Lab Abnormalities (including Chemistry, Coagulation, Hematology, and Urinalysis) | Up to 2 years plus 30 days
Change from Baseline in Vital Signs | Up to 2 years

SECONDARY OUTCOMES:
Progression-Free Survival | Until disease progression (up to 2 years)
  Progression-free survival is defined as the interval from first dose date of study drug (MMB/erlotinib) to the earlier of the first documentation of definitive disease progression or death from any cause; definitive disease progression is progression based on RECIST criteria v1.1.
Overall Survival | Until disease progression (up to 2 years)
  Overall survival is defined as the interval from first dose date of study drug (MMB/erlotinib) to death from any cause.
Overall Response Rate | Until disease progression (up to 2 years)
  Overall response rate is defined as the proportion of participants who achieve a complete response or partial response.
Pharmacokinetic (PK) Parameter: Cmax of momelotinib (MMB) | Predose and up to 24 hours postdose
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: AUCtau of momelotinib (MMB) | Predose and up to 24 hours postdose
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
PK Parameter: Cmax of Erlotinib | Predose and up to 24 hours postdose
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: AUCtau of Erlotinib | Predose and up to 24 hours postdose
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (3):
- United States (3):
  - Duarte, California
  - Palo Alto, California
  - Whittier, California

REFERENCES:
- [Derived] Padda SK, Reckamp KL, Koczywas M, Neal JW, Kawashima J, Kong S, Huang DB, Kowalski M, Wakelee HA. A phase 1b study of erlotinib and momelotinib for the treatment of EGFR-mutated, tyrosine kinase inhibitor-naive metastatic non-small cell lung cancer. Cancer Chemother Pharmacol. 2022 Jan;89(1):105-115. doi: 10.1007/s00280-021-04369-0. Epub 2021 Nov 13. PMID 34773474